CLINICAL TRIAL: NCT03515369
Title: Effect of Babaodan in Preventing Tumor Recurrence After Hepatectomy for Hepatocellular Carcinoma: a Multicenter, Randomized, Placebo-controlled, Double-blind Trial
Brief Title: Effect of Babaodan on Tumor Recurrence After Curative Resection of Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); Sun Yat-sen University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Military Medical University (Other); Xiamen Traditional Chinese Medicine Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Shen Feng, Vice President, Professor and Chief Surgeon; Member-at-large of International Hepato-Pancreato-Biliary Association (IHPBA); Secretary of Asia-Pacific Hepato-Pancreato-Biliary Association (A-PHPBA), Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EHBHKY2017-01-016
Record Dates: First submitted 2018-04-11; First posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Hepatocellular Carcinoma; Tumor Recurrence
Keywords: hepatocellular carcinoma; tumor recurrence; adjuvant therapy; traditional Chinese medicine
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepatectomy plus Babaodan (Experimental): Surgical removal of all lesions and take Babaodan oral capsule after operation
  Interventions: Drug: Babaodan oral capsule
- Hepatectomy plus Placebo (Placebo Comparator): Surgical removal of all lesions and take Placebo oral capsule after operation
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Babaodan oral capsule — On the basis of conventional liver protecting treatment, take Babaodan oral capsule within 4 weeks after curative resection. Take two capsules three times daily, two months as a course of treatment and the maximum of eighteen courses, until the recurrence of tumor or death of patients (non tumor related death), or the termination of research.
  Other Names: Conventional liver protecting treatment
  Arms: Hepatectomy plus Babaodan
Drug: Placebo oral capsule — On the basis of conventional liver protecting treatment, take Placebo oral capsule began within 4 weeks after curative resection. Take two capsules three times daily, two months as a course of treatment and the maximum of eighteen courses, until the recurrence of tumor or death of patients (non tumor related death), or the termination of research.
  Other Names: Conventional liver protecting treatment
  Arms: Hepatectomy plus Placebo

SUMMARY:
The aim of this study is to evaluate the effect of traditional Chinese medicine Babaodan on tumor recurrence of hepatocellular carcinoma after curative resection, as well as the safety of this treatment

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common malignancy and third leading cause of cancer-related mortality worldwide. Partial hepatectomy and liver transplantation are potential curative treatments for selected patients with HCC. Unfortunately, long-term surgical outcomes remain unsatisfactory due to high tumor recurrence rates, which has been reported to 40%-70%.

There are few methods for the prevention of HCC recurrence following curative-intent therapy, and no standard treatment has been established so far for recurrent tumor. The effective prevention of recurrence is the key to improve the management of this fatal malignancy. The protective role of transarterial chemoembolization (TACE) has been confirmed in advanced HCC, but the value of it as an adjuvant therapy is still controversial, which is mainly reflected in the inconsistent conclusions of the randomized controlled trials and the retrospective studies. Most prospective studies demonstrated that TACE was not effective or even harmful to postoperative tumor recurrence. Lai et al used combination therapy (lipiodol, cisplatin and epirubicin) as an adjuvant method for HCC patients after hepatectomy, and showed that the 3-year overall survival rate did not improve (66% vs. 65%), and the 3-year disease-free survival rate even decreased (18% vs. 48%) for the treatment group compared with the control group. However, retrospective studies indicate that postoperative adjuvant TACE is effective in preventing recurrence.

Immunotherapy shows its potential anti-tumor value, but its exact effect still needs further confirmation and the treatment standards is still uncertain. Compared with other solid tumors, liver cancer often has a background of hepatitis B virus (HBV) infection, so immunotherapy (such as thymosin, interferon) theoretically can simultaneously enhance the anti-tumor and anti HBV immunity, and even reduce tumor recurrence. Studies have reported that interferon treatment can improve the disease-free survival and overall survival of selected patients. Oral nucleoside antiviral drugs can improve the disease-free survival of HCC, because the hepatitis activity affects prognosis. But, the above results still need to be verified by large sample clinical trials.

Babaodan, a mixed powder of traditional Chinese medicine containing eight constituents, including natural calculus bovis, snake gall, antelope horn, pearl, musk, radix notoginseng and so on. The formula of Babaodan was protected by Chinese Food and Drug Administration. It has been widely used as a complementary and alternative medicine to treat chronic liver diseases, mitigate the side effects and enhance the efficacy of chemotherapeutic drugs, and promote cellular immunity. Lei et al reported that Babaodan can ameliorate liver injury and fibrosis in rat hepatic fibrosis model induced by diethylnitrosamine, and have no obvious side effect in normal rat livers. They also found that Babaodan did not influence the absorption of lipopolysaccharide (LPS) in liver by analysing serum from portal vein. Meanwhile, the results illustrated Babaodan can inhibit LPS-induced HSCs activation and proliferation in vitro through TLR4/NF-κB and TLR4/ERK signaling pathway, respectively. Upon these results, Babaodan may be a novel therapeutic choice for hepatic fibrosis. It also has been reported to have an effect of inhibiting the occurrence and development of HCC. However, the effect of Babaodan in preventing tumor recurrence is unclear.

In view of this, the investigators aim to implement a randomized controlled trial to assess whether oral Babaodan adjuvant therapy can effectively prevent tumor recurrence after curative resection for HCC patients, improve the quality of life, and evaluate the short-term and long-term safety of this drug.

ELIGIBILITY:
Inclusion criteria：

1. age ≥18 years and ≤75 years
2. male or female patients
3. tumor of BCLC A or B stage (≤3 nodules), and was assessed to be curative resected
4. hepatocellular carcinoma confirmed by postoperative pathology, received R0 resection
5. without tumor thrombus
6. without extrahepatic metastasis
7. KPS score ≥80
8. Child-Pugh A liver function
9. the expected postoperative survival time ≥12 weeks
10. the latest laboratory tests met the following requirements before entering the group: 1) hemoglobin ≥8.5g/dl; 2) neutrophils count ≥1,000/mm3; 3) platelet count ≥50,000/ul; 4) total bilirubin ≤2 upper limit of normal; 5) ALT and AST ≤3 upper limit of normal; 6) serum urea nitrogen and creatinine ≤1.5 upper limit of normal
11. agree to sign the informed consent

Exclusion criteria：

1. >3 tumor nodules
2. history of HCC
3. history of other tumors, except: 1) in situ carcinoma of cervix; 2) treated basal cell carcinoma; 3) superficial bladder cancer (Ta、Tis and T1); 4) any cancer that received radical treatment more than 3 years
4. with serious diseases of heart, brain, lung, kidney and blood system
5. received preoperative anti-cancer treatment
6. received radiotherapy or chemotherapy during the operation
7. pregnant or lactating women
8. receiving other clinical trials
9. history of allogeneic organ transplantation
10. patients known or suspected to be allergic to Babaodan, have allergy history of biological agents, have allergic constitution or being allergic
11. patients with hemorrhagic tendency or history of gastrointestinal bleeding within 30 days; severe esophageal varices or have history of esophageal variceal hemorrhage
12. cannot take medicine orally
13. have HIV infection or AIDS related diseases
14. have a history of mental illness or behavioral abnormality, which is assessed not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3-year
  the proportion of individuals who didn't have tumor recurrence and still alive 3 years after hepatectomy

SECONDARY OUTCOMES:
disease free survival | assessed up to 5 years
  the time from hepatectomy until tumor recurrence, death or the last follow-up time
overall survival | assessed up to 5 years
  the time from hepatectomy until death or the last follow-up time
EORTC QLQ-C30 | through study completion, an average of 3 year
  a questionnaire developed to assess the quality of life of cancer patients

OTHER OUTCOMES:
safety and tolerability | through study completion, an average of 3 year
  incidence of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, MD, PhD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided